CLINICAL TRIAL: NCT01925131
Title: S1312, A Phase I Study of Inotuzumab Ozogamicin (NSC-772518) in Combination With CVP (Cyclophosphamide, Vincristine, Prednisone) for Patients With Relapsed/Refractory CD22-Positive Acute Leukemia (Including B-ALL, Mixed Phenotypic Leukemia, and Burkitt's Leukemia)
Brief Title: S1312, Inotuzumab Ozogamicin and Combination Chemotherapy in Treating Patients With Relapsed or Refractory Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: S1312; NCI-2013-01368 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1312 (Other: SWOG); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2022-04-06 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Acute Leukemias of Ambiguous Lineage; B-cell Adult Acute Lymphoblastic Leukemia; Philadelphia Chromosome Positive Adult Precursor Acute Lymphoblastic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Cyclophosphamide; Vincristine; Prednisone; Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment (combination chemotherapy and inotuzumab ozogamicin) - Dose Level 1 (Experimental): Combination chemotherapy and inotuzumab ozogamicin - Dose level 1 Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and 0.4 mg/m2 inotuzumab ozogamicin IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: vincristine sulfate; Drug: prednisone; Biological: inotuzumab ozogamicin; Other: laboratory biomarker analysis
- Treatment (combination chemotherapy and inotuzumab ozogamicin) - Dose Level 2 (Experimental): Combination chemotherapy and inotuzumab ozogamicin - Dose level 2 Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.6 mg/m2 on day 1 and 0.4 mg/m2 on day 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: vincristine sulfate; Drug: prednisone; Biological: inotuzumab ozogamicin; Other: laboratory biomarker analysis
- Treatment (combination chemotherapy and inotuzumab ozogamicin) - Dose Level 3 (Experimental): Combination chemotherapy and inotuzumab ozogamicin - Dose level 3 Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.4 mg/m2 on day 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: vincristine sulfate; Drug: prednisone; Biological: inotuzumab ozogamicin; Other: laboratory biomarker analysis
- Treatment (combination chemotherapy and inotuzumab ozogamicin) - Dose Level 4 (Experimental): Combination chemotherapy and inotuzumab ozogamicin - Dose level 4 Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.4 mg/m2 on days 8 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: vincristine sulfate; Drug: prednisone; Biological: inotuzumab ozogamicin; Other: laboratory biomarker analysis
- Treatment (combination chemotherapy and inotuzumab ozogamicin) - Dose Level 5 (Experimental): Combination chemotherapy and inotuzumab ozogamicin - Dose level 5 Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.5 mg/m2 on days 8 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: vincristine sulfate; Drug: prednisone; Biological: inotuzumab ozogamicin; Other: laboratory biomarker analysis
- Treatment (combination chemotherapy and inotuzumab ozogamicin) - MTD (Experimental): Combination chemotherapy and inotuzumab ozogamicin - Maximum Tolerated Dose Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.5 mg/m2 on days 8 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: vincristine sulfate; Drug: prednisone; Biological: inotuzumab ozogamicin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Biological: inotuzumab ozogamicin — Given IV
  Other Names: CMC-544
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of inotuzumab ozogamicin when given together with combination chemotherapy in treating patients with relapsed or refractory acute leukemia. Immunotoxins, such as inotuzumab ozogamicin, can find cancer cells that express cluster of differentiation (CD)22 and kill them without harming normal cells. Drugs used in chemotherapy, such as cyclophosphamide, vincristine sulfate, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving inotuzumab ozogamicin together with combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of inotuzumab ozogamicin in combination with cyclophosphamide, vincristine (vincristine sulfate) and prednisone (CVP) and to determine the maximum tolerated dose (MTD) of inotuzumab ozogamicin in this regimen for patients with relapsed or refractory CD22+ acute leukemia (B-cell acute lymphoblastic leukemia [B-ALL], mixed phenotype, and Burkitt's).

SECONDARY OBJECTIVES:

I. To estimate the preliminary activity (response rate: complete remission [CR] + complete remission with incomplete count recovery [CRi]) of this combination in the expansion cohort.

II. To estimate the frequency and severity of toxicities of this combination in this patient population.

OUTLINE: This is a dose-escalation study of inotuzumab ozogamicin.

Patients receive cyclophosphamide intravenously (IV) on day 1, vincristine sulfate IV on day 1, prednisone orally (PO) on days 1-5, and inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 1 year, every 3 months for 1 year, and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of relapsed or refractory CD22-positive acute leukemia including B-ALL, mixed phenotype leukemia (biphenotypic), or Burkitt's leukemia based on World Health Organization (WHO) classification; patients with bilineal leukemia are excluded
* Patients must have evidence of acute leukemia in their peripheral blood or bone marrow; patients must have >= 5% blasts in the peripheral blood or bone marrow within 14 days prior to registration; at least >= 20% of those blasts must be CD22-positive (surface) based on local immunophenotyping and histopathology
* Patients must be refractory or have relapsed following prior induction therapy; a standard induction regimen is defined as any program of treatment that includes vincristine and prednisone or dexamethasone, cytarabine/anthracycline, or high dose cytarabine
* For sites with the B1931022 pharmaceutical trial open, precursor B-cell ALL patients from that site may be eligible for S1312 providing they meet the following criteria:

  * Patient is in second salvage or more; OR
  * Patient was treated on the standard of care arm of B1931022 and failed therapy
* Patients may have received prior allogeneic transplant or autologous transplant; however, patients with prior allogeneic bone marrow transplant will be eligible only if both of the following conditions are met:

  * The transplant must have been performed >= 90 days prior to registration
  * The patient must not have >= grade 2 acute graft versus host disease (GvHD) or either moderate or severe limited chronic GvHD within 14 days prior to registration
* Patients known to have Philadelphia chromosome positive (Ph+) ALL must have either failed treatment or been intolerant to treatment with at least two second or third generation tyrosine kinase inhibitors
* Patients must not have received prior treatment with inotuzumab ozogamicin; previous treatment with other anti-CD22 antibodies must have been completed at least 90 days prior to registration
* Patients must have Zubrod performance status 0-2
* Patients must not have received any chemotherapy, investigational agents, or undergone major surgery within 14 days prior to registration with the following exceptions:

  * Monoclonal antibodies must not have been received for 1 week prior to registration
  * Chimeric antigen receptor (CAR) T-cells must not have been received for 28 days prior to registration.
  * Steroids, hydroxyurea, vincristine, 6-mercaptopurine, methotrexate, thioguanine and intrathecal chemotherapy are permitted within any time frame prior to registration. FDA-approved TKIs may also be administered until 1 day prior to start of study therapy (C1, D1).
  * All drug-related toxicities must have resolved to =< grade 2
* Patients must not have a systemic bacterial, fungal, or viral infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement despite appropriate antibiotics or other treatment)
* Patients must not have any other serious concurrent disease or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that would put the patient at undue risk of undergoing therapy
* Patients must not have active central nervous system (CNS) involvement (by clinical evaluation); patients with previous documented history of CNS involvement of acute leukemia, or with clinical signs or symptoms consistent with CNS involvement of acute leukemia, must have a lumbar puncture which is negative for CNS involvement of acute leukemia; the lumbar puncture must be completed within 14 days prior to registration; patients with no previous history of documented CNS involvement and with no clinical signs or symptoms consistent with CNS involvement are not required to have completed a lumbar puncture before registration; note that treatment with intrathecal therapy is recommended during protocol treatment but CNS analysis during treatment is not required
* Patients must have a peripheral blast count < 25,000/uL within 2 days prior to registration; (treatment with hydroxyurea and steroids is permitted to bring the countdown)
* Patients must have serum creatinine =< 2 x institutional upper limits of normal (IULN) within 7 days prior to registration
* Patients must have bilirubin =< 2 x IULN within 7 days prior to registration (unless the bilirubin is primarily unconjugated)
* Patients must have < grade 2 neuropathy (sensory/motor) within 7 days prior to registration
* Patients must have serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 2.5 x IULN within 7 days prior to registration
* Patients with a history of a serious allergic or anaphylactic reaction to humanized monoclonal antibodies are not eligible
* Patients must not have a history of chronic or active hepatitis B or C infection; patients must have negative hepatitis B and C serologies performed within 28 days prior to registration
* Patients must not have evidence or history of veno-occlusive disease or sinusoidal obstruction syndrome
* Patients must not have a cardiac ejection fraction < 45% or the presence of New York Heart Association stage III or IV heart failure within 14 days prior to registration; either echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA) may be used to determine ejection fraction
* Patients must not have a myocardial infarction within 6 months prior to registration
* Patients must not have a history of clinically significant arrhythmia, prolonged corrected QT (QTc) interval, or unexplained syncope not thought to be vasovagal in nature within 6 months prior to registration
* Patients must not have a screening corrected QT using Fridericia's formula (QTcF) interval > 500 milliseconds (by Fridericia calculation) based on the average of triplicate electrocardiogram (EKG) performed within 7 days prior to registration; note that triplicate EKG is required at other timepoints
* Patients must not have a history of chronic liver disease (or cirrhosis)
* Patients who are known to be human immunodeficiency virus (HIV)+ are eligible providing they meet all of the following additional criteria within 28 days prior to registration:

  * CD4+ cells >= 350/mm^3 (nadir)
  * Viral load of < 50 copies HIV messenger ribonucleic acid (mRNA)/mm^3 if on combination antiretroviral therapy (cART) or < 25,000 copies HIV mRNA if not on cART
  * No zidovudine or stavudine as part of cART Patients who are HIV+ and do not meet all of these criteria are not eligible for this study
* Patients with evidence of extramedullary disease at diagnosis will have computed tomography (CT) scan of the chest, abdomen and pelvis to obtain baseline values within 28 days prior to registration
* Patients must have complete history and physical examination within 28 days prior to registration
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Prior malignancy other than acute leukemia is allowed, provided it is in remission and there is no plan to treat the malignancy at the time of registration
* Pretreatment cytogenetics must be performed on all patients; collection of pretreatment specimens must be completed within 14 days prior to registration to S1312; specimens must be submitted to the site's preferred Clinical Laboratory Improvement Amendments (CLIA)-approved cytogenetics laboratory; reports of the results must be submitted as described; note that cytogenetics are required at other time points
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Patients planning to enroll in this study must first have a slot reserved in advance of the registration; all site staff will use OPEN to create a slot reservation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, Principal Investigator — SWOG Cancer Research Network
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of Rochester, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ben Taub General Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were a total of 50 participants enrolled. However, two were deemed ineligible due to inadequate liver function and did not start protocol treatment, leaving 48 eligible participants.
Groups:
- CVP + Inotuzumab Dose Level 1: Combination chemotherapy and inotuzumab ozogamicin - Dose level 1
  Patients receive 750 mg/m2 cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and 0.4 mg/m2 inotuzumab ozogamicin IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab Dose Level 2: Combination chemotherapy and inotuzumab ozogamicin - Dose level 2
  Patients receive 750 mg/m2 cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.6 mg/m2 on day 1 and 0.4 mg/m2 on day 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab Dose Level 3: Combination chemotherapy and inotuzumab ozogamicin - Dose level 3
  Patients receive 750 mg/m2 cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.4 mg/m2 on day 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab Dose Level 4: Combination chemotherapy and inotuzumab ozogamicin - Dose level 4
  Patients receive 750 mg/m2 cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.4 mg/m2 on days 8 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab Dose Level 5: Combination chemotherapy and inotuzumab ozogamicin - Dose level 5
  Patients receive 750 mg/m2 cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.5 mg/m2 on days 8 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab MTD (Expansion Cohort): Combination chemotherapy and inotuzumab ozogamicin - Maximum Tolerated Dose (Expansion Cohort)
  Patients receive 750 mg/m2 cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.5 mg/m2 on days 8 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | CVP + Inotuzumab Dose Level 1 | CVP + Inotuzumab Dose Level 2 | CVP + Inotuzumab Dose Level 3 | CVP + Inotuzumab Dose Level 4 | CVP + Inotuzumab Dose Level 5 | CVP + Inotuzumab MTD (Expansion Cohort)
Started | 5 | 4 | 10 | 5 | 11 | 13
Completed | 0 | 2 | 1 | 0 | 0 | 3
Not Completed | 5 | 2 | 9 | 5 | 11 | 10
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progression/Relapse | 1 | 1 | 4 | 0 | 0 | 1
Not completed — Patient Refusal | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 1 | 3
Not completed — Other - Not Protocol Specified | 3 | 1 | 2 | 5 | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- CVP + Inotuzumab Dose Level 1: Combination chemotherapy and inotuzumab ozogamicin � Dose level 1
  Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and 0.4 mg/m2 inotuzumab ozogamicin IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab Dose Level 2: Combination chemotherapy and inotuzumab ozogamicin - Dose level 2
  Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.6 mg/m2 on day 1 and 0.4 mg/m2 on day 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab Dose Level 3: Combination chemotherapy and inotuzumab ozogamicin - Dose level 3
  Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.4 mg/m2 on day 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab Dose Level 4: Combination chemotherapy and inotuzumab ozogamicin - Dose level 4
  Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.4 mg/m2 on days 8 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab Dose Level 5: Combination chemotherapy and inotuzumab ozogamicin - Dose level 5
  Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.5 mg/m2 on days 8 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- CVP + Inotuzumab MTD: Combination chemotherapy and inotuzumab ozogamicin - Maximum Tolerated Dose
  Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour at 0.8 mg/m2 on day 1 and 0.5 mg/m2 on days 8 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | CVP + Inotuzumab Dose Level 1 | CVP + Inotuzumab Dose Level 2 | CVP + Inotuzumab Dose Level 3 | CVP + Inotuzumab Dose Level 4 | CVP + Inotuzumab Dose Level 5 | CVP + Inotuzumab MTD | Total
Number analyzed (Participants) | 5 | 4 | 10 | 5 | 11 | 13 | 48
Age, Continuous [Median (Full Range); unit: years] | 48.8 [22.3 to 73.7] | 42.3 [20.6 to 56.4] | 42.8 [22.4 to 75.3] | 49.6 [33.0 to 50.1] | 37.9 [25.0 to 58.7] | 43.5 [21.6 to 79.8] | 43 [20.6 to 79.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 4 | 2 | 5 | 5 | 21
  Male | 4 | 0 | 6 | 3 | 6 | 8 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 4 | 3 | 3 | 16
  Not Hispanic or Latino | 3 | 2 | 7 | 1 | 6 | 9 | 28
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 1 | 0 | 5
  White | 4 | 3 | 6 | 5 | 7 | 8 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: MTD of Inotuzumab Ozogamicin With CVP for Patients With Relapsed or Refractory CD22+ Acute Leukemia
Description: To determine the maximum tolerated dose (MTD) of inotuzumab ozogamicin in this regimen for patients with relapsed or refractory CD22+ acute leukemia (B-cell acute lymphoblastic leukemia [B-ALL], mixed phenotype, and Burkitt's). The MTD is defined as the highest dose studied in which the incidence of dose-limiting toxicities is < 33% using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.
Time Frame: 28 days
Population: Includes eligible patients who received treatment among all arms.
Measure: Number; unit: mg/m^2
Groups:
- CVP + Inotuzumab: Combination chemotherapy and inotuzumab ozogamicin
  Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | CVP + Inotuzumab
Number analyzed (Participants) | 48
mg/m^2
  Day 1 Dose | 0.8
  Day 8 Dose | 0.5
  Day 15 Dose | 0.5

2. Secondary Outcome: Response Rate (CR+CRi) Among Expansion Cohort
Description: The response rate (CR + CRi) is defined as the rate of complete remission (CR) + complete remission with incomplete count recovery (CRi). Complete remission (CR) is defined as < 5% marrow aspirate blasts, neutrophils ≥ 1000/uL, platelets > 100,000/uL, no blasts in peripheral blood, and C1 Extramedullary disease status. C1 Extramedullary disease status is characterized by complete disappearance of all measurable and non-measurable extramedullary disease with the exception of lesions for which the following must be true: for participants with at least one measurable lesion, all lesions must have reduced by 75% in sum of products of greatest diameters (SPD), have no new lesions, and the spleen and other previously enlarged organs must have regressed in size. Complete remission with incomplete platelet recovery (CRi) is defined the same as CR, except absolute neutrophil count may be <1000/uL and/or platelet count may be ≤ 100,000/uL.
Time Frame: Up to 3 years
Population: MTD arm only, including eligible patients who received treatment and were evaluable for response
Measure: Number; unit: percentage of participants
Arm/Group | CVP + Inotuzumab MTD
Number analyzed (Participants) | 12
percentage of participants | 83.33

3. Secondary Outcome: Frequency and Severity of Toxicities
Description: Number of participants with Grade 3-5 adverse events that are possibly, probably or definitely related to study drug are reported by given type of adverse event.
Time Frame: Up to 3 years
Population: Eligible participants who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- CVP + Inotuzumab Dose Level 1: Combination chemotherapy and inotuzumab ozogamicin - Dose level 1
  Patients receive cyclophosphamide IV on day 1, vincristine sulfate IV on day 1, prednisone PO on days 1-5, and 0.4 mg/m2 inotuzumab ozogamicin IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | CVP + Inotuzumab Dose Level 1 | CVP + Inotuzumab Dose Level 2 | CVP + Inotuzumab Dose Level 3 | CVP + Inotuzumab Dose Level 4 | CVP + Inotuzumab Dose Level 5 | CVP + Inotuzumab MTD
Number analyzed (Participants) | 5 | 4 | 10 | 5 | 11 | 13
Participants
  Anemia | 2 | 2 | 7 | 3 | 5 | 5
  Ascites | 0 | 0 | 0 | 0 | 1 | 1
  Dysphagia | 0 | 0 | 1 | 0 | 0 | 0
  Encephalopathy | 0 | 0 | 1 | 0 | 0 | 0
  Enterocolitis | 0 | 0 | 0 | 0 | 1 | 0
  Fatigue | 0 | 0 | 1 | 0 | 0 | 1
  Febrile neutropenia | 0 | 2 | 2 | 3 | 1 | 7
  Fever | 1 | 1 | 1 | 0 | 0 | 1
  Gastric hemorrhage | 2 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Other, specify | 0 | 1 | 0 | 0 | 0 | 0
  Headache | 0 | 1 | 0 | 0 | 0 | 0
  Hyperglycemia | 0 | 0 | 4 | 4 | 2 | 0
  Hypertension | 0 | 0 | 1 | 1 | 0 | 1
  Hypoalbuminemia | 0 | 0 | 1 | 0 | 0 | 0
  Hypocalcemia | 0 | 0 | 1 | 0 | 0 | 0
  Hypokalemia | 0 | 0 | 0 | 1 | 0 | 0
  Infections and infestations - Other, specify | 0 | 0 | 0 | 0 | 1 | 4
  Intracranial hemorrhage | 1 | 0 | 0 | 0 | 0 | 0
  Lipase increased | 0 | 0 | 0 | 0 | 0 | 1
  Lung infection | 0 | 0 | 0 | 2 | 0 | 0
  Lymphocyte count decreased | 2 | 1 | 3 | 3 | 6 | 6
  Mucositis oral | 0 | 0 | 1 | 0 | 0 | 1
  Neutrophil count decreased | 3 | 3 | 9 | 4 | 8 | 8
  Platelet count decreased | 2 | 2 | 7 | 4 | 5 | 10
  Renal and urinary disorders - Other, specify | 0 | 0 | 0 | 0 | 0 | 1
  Sepsis | 0 | 0 | 0 | 0 | 0 | 2
  Skin infection | 0 | 0 | 1 | 0 | 0 | 0
  White blood cell decreased | 3 | 4 | 10 | 5 | 7 | 9

ADVERSE EVENTS:
Time Frame: Up to 3 years post registration
Description: All adverse events, regardless of attribution and grade, are reported.
Arm/Group | CVP + Inotuzumab Dose Level 1 | CVP + Inotuzumab Dose Level 2 | CVP + Inotuzumab Dose Level 3 | CVP + Inotuzumab Dose Level 4 | CVP + Inotuzumab Dose Level 5 | CVP + Inotuzumab MTD
All-Cause Mortality (participants affected / at risk) | 4/5 | 3/4 | 9/10 | 5/5 | 9/11 | 8/13
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/4 | 4/10 | 1/5 | 1/11 | 11/13
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 10/10 | 5/5 | 11/11 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVP + Inotuzumab Dose Level 1 (N=5) | CVP + Inotuzumab Dose Level 2 (N=4) | CVP + Inotuzumab Dose Level 3 (N=10) | CVP + Inotuzumab Dose Level 4 (N=5) | CVP + Inotuzumab Dose Level 5 (N=11) | CVP + Inotuzumab MTD (N=13)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Edema face (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Fever (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Infections and infestations-Other (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 5
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Investigations-Other (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Nervous system disorders-Other (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal and urinary disorders-Other (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CVP + Inotuzumab Dose Level 1 (N=5) | CVP + Inotuzumab Dose Level 2 (N=4) | CVP + Inotuzumab Dose Level 3 (N=10) | CVP + Inotuzumab Dose Level 4 (N=5) | CVP + Inotuzumab Dose Level 5 (N=11) | CVP + Inotuzumab MTD (N=13)
Anemia (Blood and lymphatic system disorders) | 3 | 3 | 9 | 5 | 10 | 9
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3 | 2 | 8
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac disorders-Other (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 1 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 6 | 4 | 4 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ear and labyrinth disorders-Other (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blurred vision (Eye disorders) | 1 | 1 | 0 | 2 | 1 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 1 | 0 | 0 | 0 | 0
Eye disorders-Other (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Watering eyes (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 7
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 3 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 0 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 4
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 5 | 3 | 2 | 6
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 3
Chills (General disorders) | 1 | 0 | 1 | 1 | 1 | 8
Edema face (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 1 | 6 | 3 | 2 | 4
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 3 | 1 | 5 | 5
Fever (General disorders) | 3 | 2 | 2 | 2 | 1 | 4
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
General disorders and admin site conditions - Other (General disorders) | 0 | 0 | 0 | 0 | 0 | 4
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 2 | 1 | 2
Pain (General disorders) | 2 | 1 | 4 | 1 | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations-Other (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 5
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 2 | 3 | 5 | 6
Alkaline phosphatase increased (Investigations) | 3 | 1 | 4 | 4 | 7 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 2 | 3 | 7 | 2
Blood bilirubin increased (Investigations) | 0 | 2 | 3 | 1 | 1 | 5
Cholesterol high (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0
Fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Investigations-Other (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 2 | 3 | 3 | 7 | 6
Neutrophil count decreased (Investigations) | 3 | 3 | 9 | 4 | 10 | 9
Platelet count decreased (Investigations) | 3 | 3 | 8 | 5 | 10 | 10
Weight gain (Investigations) | 0 | 1 | 1 | 1 | 1 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
White blood cell decreased (Investigations) | 3 | 4 | 10 | 5 | 10 | 10
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 2 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 1 | 5 | 4 | 7 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2 | 6 | 4 | 9 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 2 | 3 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 3 | 8 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2 | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 3 | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2 | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 2 | 3 | 4
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 1 | 0 | 3
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Facial muscle weakness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 3 | 3 | 7
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 2 | 2 | 2
Memory impairment (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1
Nervous system disorders-Other (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 2 | 1 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 3 | 3 | 6
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 2 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 3 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 3 | 1 | 2 | 0
Confusion (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 2 | 3 | 2
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Psychiatric disorders-Other (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 2
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 1
Renal and urinary disorders-Other (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1 | 2 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 3 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 4 | 3 | 5 | 3
Hypotension (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 3
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT01925131/Prot_SAP_ICF_000.pdf